CLINICAL TRIAL: NCT00956020
Title: Evaluation of the Mechanism of Action of Platelet Rich Fibrin Matrix (PRFM) in Producing Skin Volume Augmentation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The New York Eye & Ear Infirmary (Other)
Responsible Party: Principal Investigator, Anthony P. Sclafani, Director of Facial Plastic Surgery, The New York Eye & Ear Infirmary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-01
Record Dates: First submitted 2009-08-10; First posted 2009-08-11 (Estimated); Results first posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Aging
Keywords: platelet rich plasma; fibrin matrix; dermal filler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies over a period from 30 minutes to 12 weeks after treatment.
  Interventions: Biological: Platelet rich fibrin matrix

INTERVENTIONS:
Biological: Platelet rich fibrin matrix — Single treatment with platelet rich fibrin matrix
  Other Names: Selphyl

SUMMARY:
Autologous platelet rich fibrin matrix will release growth factors which could increase the production of dermal proteins or affect the vascularity and status of neighboring tissues. This study is designed to evaluate the histologic and biochemical effect of injection of platelet rich fibrin matrix into the skin.

DETAILED DESCRIPTION:
Subjects will be treated with platelet rich fibrin matrix into the skin of the inner aspect of the upper arm. Injected areas will be monitored clinically and will also undergo biopsies between 30 minutes and 12 weeks after treatment. Specimen of treated areas will undergo histologic and biochemical analysis and comparison to standard laboratory control specimen of untreated skin.

ELIGIBILITY:
Inclusion Criteria:

* 25 and 75 years of age

Exclusion Criteria:

* collagen vascular disorders
* autoimmune diseases
* signs or history of impaired wound healing
* shall not have had any infectious or inflammatory processes at the treatment sites within the prior 6 months

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2011-02 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Sclafani, MD, Principal Investigator — The NY Eye & Ear Infirmary
Locations (1):
- The NY Eye & Ear Infirmary, New York, New York, United States

REFERENCES:
- [Result] Sclafani AP, McCormick SA. Induction of dermal collagenesis, angiogenesis, and adipogenesis in human skin by injection of platelet-rich fibrin matrix. Arch Facial Plast Surg. 2012 Mar-Apr;14(2):132-6. doi: 10.1001/archfacial.2011.784. Epub 2011 Oct 17. PMID 22006233

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies over a 12 week period.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Period: Overall Study
Arm/Group | Treatment
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Collagen and Cellularity 30 Minutes After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal collagen (as determined by the number of specimen which had greater than 25% new collagen deposition per high powered field) 30 minutes after treatment with platelet rich fibrin matrix will be reported. The results were characterize the general qualitative changes and time frame for the effects of treatment.
Time Frame: 30 minutes after treatment
Population: Each participant will undergo biopsy of skin treated with platelet rich fibrin matrix, at 30 minutes after treatment.
Measure: Number; unit: %specimen with >25%new collagen/HPF
Units Other Than Participants: skin biopsy specimen
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies over a period from 30 minutes to 12 weeks after treatment.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 4
Number analyzed (skin biopsy specimen) | 4
%specimen with >25%new collagen/HPF | 0

2. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Collagen and Cellularity 1 Week After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal collagen (as determined by the number of specimen which had greater than 25% new collagen deposition per high powered field) 1 week after treatment with platelet rich fibrin matrix will be reported. The results were characterize the general qualitative changes and time frame for the effects of treatment.
Time Frame: 1 week after treatment
Population: Each participant will undergo biopsy of skin treated with platelet rich fibrin matrix, at 1 week after treatment.
Measure: Number; unit: %specimen with >25%new collagen/HPF
Units Other Than Participants: Skin biopsy specimen
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 1 week after treatment.
  Platelet rich fibrin matrix: Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 3
Number analyzed (Skin biopsy specimen) | 3
%specimen with >25%new collagen/HPF | 100

3. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Collagen and Cellularity 2 Weeks After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal collagen (as determined by the number of specimen which had greater than 25% new collagen deposition per high powered field) 2 weeks after treatment with platelet rich fibrin matrix will be reported. The results were characterize the general qualitative changes and time frame for the effects of treatment.
Time Frame: 2 weeks after treatment
Population: Each participant will undergo biopsy of skin treated with platelet rich fibrin matrix, at 2 weeks after treatment.
Measure: Number; unit: %specimen with >25%new collagen/HPF
Units Other Than Participants: skin biopsy specimen
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 2 weeks after treatment.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 2
Number analyzed (skin biopsy specimen) | 2
%specimen with >25%new collagen/HPF | 100

4. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Collagen and Cellularity 6 Weeks After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal collagen (as determined by the number of specimen which had greater than 25% new collagen deposition per high powered field) 6 weeks after treatment with platelet rich fibrin matrix will be reported. The results were characterize the general qualitative changes and time frame for the effects of treatment.
Time Frame: 6 weeks after treatment
Population: Each participant will undergo biopsy of skin treated with platelet rich fibrin matrix, at 6 weeks after treatment.
Measure: Number; unit: %specimen with >25%new collagen/HPF
Units Other Than Participants: Skin biopsy specimen
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 6 weeks after treatment.
  Platelet rich fibrin matrix: Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 3
Number analyzed (Skin biopsy specimen) | 3
%specimen with >25%new collagen/HPF | 100

5. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Collagen and Cellularity 10 Weeks After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal collagen (as determined by the number of specimen which had greater than 25% new collagen deposition per high powered field) 10 weeks after treatment with platelet rich fibrin matrix will be reported. The results were characterize the general qualitative changes and time frame for the effects of treatment.
Time Frame: 10 weeks after treatment
Population: Each participant will undergo biopsy of skin treated with platelet rich fibrin matrix, at 10 weeks after treatment.
Measure: Number; unit: %specimen with >25%new collagen/HPF
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 10 weeks after treatment.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 2
%specimen with >25%new collagen/HPF | 100

6. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Collagen and Cellularity 12 Weeks After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal collagen (as determined by the number of specimen which had greater than 25% new collagen deposition per high powered field) 12 weeks after treatment with platelet rich fibrin matrix will be reported. The results were characterize the general qualitative changes and time frame for the effects of treatment.
Time Frame: 12 weeks after treatment
Population: Each participant will undergo biopsy of skin treated with platelet rich fibrin matrix, at 12 weeks after treatment.
Measure: Number; unit: %specimen with >25%new collagen/HPF
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 12 weeks after treatment.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 2
%specimen with >25%new collagen/HPF | 100

7. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Vascularity 30 Minutes After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal vascularity (as determined by the the number of specimen with greater than 5 immature capillaries per high powered field) after treatment with platelet rich fibrin matrix will be reported. Individual treated specimen were evaluated at 30 minutes after treatment, and the results used to determine the general qualitative changes and time frame for the effects of treatment.
Time Frame: 30 minutes after treatment
Population: Each participant underwent biopsy of skin treated with platelet rich fibrin matrix at 30 minutes.
Measure: Number; unit: % spec.with>5 immature capillaries/HPF
Units Other Than Participants: Skin biopsy specimen
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 30 minutes after treatment.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 4
Number analyzed (Skin biopsy specimen) | 4
% spec.with>5 immature capillaries/HPF | 0

8. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Vascularity 1 Week After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal vascularity (as determined by the the number of specimen with greater than 5 immature capillaries per high powered field) after treatment with platelet rich fibrin matrix will be reported. Individual treated specimen were evaluated at 1 week after treatment, and the results used to determine the general qualitative changes and time frame for the effects of treatment.
Time Frame: 1 week after treatment
Population: Each participant underwent biopsy of skin treated with platelet rich fibrin matrix at 1 week.
Measure: Number; unit: % spec.with>5 immature capillaries/HPF
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 1 week after treatment.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 3
% spec.with>5 immature capillaries/HPF | 100

9. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Vascularity 2 Weeks After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal vascularity (as determined by the number of specimen with greater than 5 immature capillaries per high powered field) after treatment with platelet rich fibrin matrix will be reported. Individual treated specimen were evaluated at 2 weeks after treatment, and the results used to determine the general qualitative changes and time frame for the effects of treatment.
Time Frame: 2 weeks after treatment
Population: Each participant underwent biopsy of skin treated with platelet rich fibrin matrix at 2 weeks.
Measure: Number; unit: % spec.with>5 immature capillaries/HPF
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 2 week after treatment.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 2
% spec.with>5 immature capillaries/HPF | 100

10. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Vascularity 6 Weeks After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal vascularity (as determined by the number of specimen with greater than 5 immature capillaries per high powered field) after treatment with platelet rich fibrin matrix will be reported. Individual treated specimen were evaluated at 6 weeks after treatment, and the results used to determine the general qualitative changes and time frame for the effects of treatment.
Time Frame: 6 weeks after treatment
Population: Each participant underwent biopsy of skin treated with platelet rich fibrin matrix at 6 weeks.
Measure: Number; unit: % spec.with>5 immature capillaries/HPF
Groups:
- Treatment: Skin injection with platelet rich fibrin matrix on the inner aspect of the upper arm, with biopsies 6 weeks after treatment.
  Platelet rich fibrin matrix : Single treatment with platelet rich fibrin matrix
Arm/Group | Treatment
Number analyzed (Participants) | 3
% spec.with>5 immature capillaries/HPF | 100

11. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Vascularity 10 Weeks After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal vascularity (as determined by the number of specimen with greater than 5 immature capillaries per high powered field) after treatment with platelet rich fibrin matrix will be reported. Individual treated specimen were evaluated at 10 weeks after treatment, and the results used to determine the general qualitative changes and time frame for the effects of treatment.
Time Frame: 10 weeks after treatment
Population: Each participant underwent biopsy of skin treated with platelet rich fibrin matrix at 10 weeks.
Measure: Number; unit: % spec.with>5 immature capillaries/HPF
Arm/Group | Treatment
Number analyzed (Participants) | 2
% spec.with>5 immature capillaries/HPF | 100

12. Primary Outcome: Qualitative Changes in Dermal and Sub Dermal Vascularity 12 Weeks After Treatment With Platelet Rich Fibrin Matrix
Description: Biopsy specimen will be obtained from PRFM treated skin, sectioned and stained with H&E. Qualitative differences from standard laboratory control specimen of normal untreated skin (not obtained from study participants) in dermal and sub dermal vascularity (as determined by the number of specimen with greater than 5 immature capillaries per high powered field) after treatment with platelet rich fibrin matrix will be reported. Individual treated specimen were evaluated at 12 weeks after treatment, and the results used to determine the general qualitative changes and time frame for the effects of treatment.
Time Frame: 12 weeks after treatment
Population: Each participant underwent biopsy of skin treated with platelet rich fibrin matrix at 12 weeks.
Measure: Number; unit: % spec.with>5 immature capillaries/HPF
Arm/Group | Treatment
Number analyzed (Participants) | 2
% spec.with>5 immature capillaries/HPF | 50

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No